CLINICAL TRIAL: NCT01101776
Title: Post Marketing Surveillance Study to Evaluate the Tolerability of Rebif® New Formulation in Patients With Relapsing Multiple Sclerosis in an Australian Clinical Setting
Acronym: ReNew
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 701068-522
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, relapsing; Rebif New Formulation; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon beta-1a (Rebif) — Interferon beta-1a 44 micrograms (12 MIU) given three times per week (tiw) by subcutaneous injection (SCI). Dose to be reduced to 22 micrograms (6 MIU) tiw by SCI for subjects who cannot tolerate the higher dose.
  Other Names: Rebif New Formulation

SUMMARY:
This observational multicentric study is planned to assess the tolerability of Rebif New Formulation in an Australian clinical setting by the incidence of injection site reactions (ISRs). The study will allow the comparison of tolerability data with historical data for both Rebif New and classic formulations, and will do so by using the same pre- specified preferred terms of treatment emergent adverse events as done in historical studies. In addition, the study will analyse whether interaction(s) with a nurse impacts tolerability and the impact of Rebif New Formulation on the patient's Quality of Life.

DETAILED DESCRIPTION:
The disease-modifying therapies for multiple sclerosis (MS) aim to slow down the disease process and consequent damage to central nervous system. This study is an open-label, multicentric study planned to assess the tolerability of Rebif New Formulation in an Australian clinical setting by the incidence of ISRs. A total of 100 subjects having relapsing MS across approximately 20 sites in Australia will be enrolled into the study. Subject visits will be scheduled at baseline (month 0) and months 3, 6, 9 and 12 and the data related to demographic factors, disease history, quality of life and adverse drug reactions (ADRs) will be recorded in the case report form (CRF).

OBJECTIVES

Primary Objective:

* To assess the tolerability of Rebif New Formulation in an Australian clinical setting by the incidence of ISRs

Secondary Objectives:

* Observe the number of and reasons for missed injections of Rebif New Formulation at 3, 6, 9 and 12 months
* Assess changes in quality of life [Multiple Sclerosis International Quality of Life Questionaire (MusiQoL)] at 6 and 12 months compared to baseline
* Number and type (telephone, face-to-face, written) of interactions with nurse support at 3, 6, 9 and 12 months.
* Assess relapse rate at 12 months
* Assess any differences in tolerability of Rebif New Formulation between subjects who were treatment naïve or on previous MS therapy
* Observe the proportion of subjects with dose reductions to 22 mcg as a result of tolerability

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with Multiple Sclerosis who:

  1. have experienced two or more relapses within the last 2 years. or
  2. are not tolerating their current MS therapy.
* Patients 18 years of age or over.
* Patients with Expanded Disability Status Scale (EDSS) score <6.0.
* Patients who have given informed consent to participate in the study.

Exclusion Criteria:

* Subjects with diagnosis of any other form of MS other than relapsing MS.
* Contra-indicated medical conditions for IFN beta-1a as defined in the Product Information i.e: women who are or plan to become pregnant whilst on therapy; subject with severe depressive disorders and/or suicidal ideation and; epileptic subjects with seizures not adequately controlled by treatment
* Subjects with a known hypersensitivity to natural or recombinant interferon beta, mannitol, poloxamer, methionine, sodium acetate buffer or benzyl alcohol.
* Subjects who are pregnant and/or breastfeeding.
* Subjects currently on Rebif New Formulation.
* Subjects currently experiencing a relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with MS who have experienced two or more relapses within last 2 years and to be treated with Rebif New Formulation in Australia.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence and type of injection site reactions (ISRs) | Month 3, 6, 9 and 12

SECONDARY OUTCOMES:
Number of missed injections of Rebif New Formulation since the previous visit | Month 3, 6, 9 and 12
Reasons for missed injections of Rebif New Formulation since the previous visit | Month 3, 6, 9 and 12
Changes in quality of life (MusiQoL) | Baseline visit and at Month 6 and 12
Number and type (telephone, face-to-face, written) of interactions with nurse support | Month 3, 6, 9 and 12
Relapse rate | Month 3, 6, 9 and 12.
Proportion of subjects with dose reductions to 22 mcg as a result of tolerability | Month 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sartori, Study Director — Merck Serono Australia Pty Ltd
Locations (15):
- Australia (15):
  - Merck Serono Research Site, Bruce, Australian Capital Territory
  - Merck Serono Research Site, Burwood, New South Wales
  - Merck Serono Research Site, Chatswood, New South Wales
  - Merck Serono Research Site, Orange, New South Wales
  - Merck Serono Research Site, Rozelle, New South Wales
  - Merck Serono Research Site, Woollongong, New South Wales
  - Merck Serono Research Site, Adelaide, South Australia
  - Merck Serono Research Site, Box Hill, Victoria
  - Merck Serono Research Site, Clayton, Victoria
  - Merck Serono Research Site, Fitzroy, Victoria
  - Merck Serono Research Site, Footscray, Victoria
  - Merck Serono Research Site, Geelong, Victoria
  - Merck Serono Research Site, Heidelberg, Victoria
  - Merck Serono Research Site, Nedlands, Western Australia
  - Merck Serono Research Site, Perth, Western Australia